CLINICAL TRIAL: NCT07185763
Title: Feasibility and Outcomes of Nano-Learning for Improving Compliance With Physical and Nutritional Guidelines and Reducing Late-Life Depression Among Older Adults With Sarcopenia in a Rural Province
Brief Title: Nano-Learning for Improving Compliance Among Older Adults With Sarcopenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, assistant professor, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 7/9/2025
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Learning; Lack of (Specific); Depression; Older Adults; Sarcopenia
MeSH Terms: conditions — Depression; Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): • Recruitment was conducted through face-to-face interviews in the clinic's waiting areas by the research team. These initial meetings, lasting approximately 20-30 minutes per participant, were essential for building rapport, obtaining anthropometric and other objective data, and ensuring informed consent. During the interview, the researchers explained the purpose and procedures of the study in detail, collected participants' mobile phone numbers, and administered the baseline (pretest) assessment using the study tools.
  Interventions: Behavioral: Nano-Learning interventional program
- control (No Intervention): they will be exposed only to the routine care provided by the nursing homes.

INTERVENTIONS:
Behavioral: Nano-Learning interventional program — AI-based Nano-learning videos involves designing ultra-short, single-focus lessons (not exceeding 2 minutes). Each session was delivered in form of some videos.
  Arms: interventional group

SUMMARY:
Empirical evidence suggests that the use of short videos is associated with decreased feelings of loneliness and social isolation, thereby reducing depression among older adults . Platforms that allow users to showcase aspects of their own lives also serve as a significant avenue for achieving "happiness in old age" and enhancing social interactions with acquaintances . Therefore, this study aims to provide robust evidence on the effectiveness of nano-learning interventions, particularly in the context of sarcopenia, where addressing physical and psychological well-being has become increasingly critical among this cohort.

DETAILED DESCRIPTION:
Nanolearning is an innovative pedagogical strategy that delivers content in highly focused, ultra-short learning experiences, often lasting less than two minutes, aimed at teaching a single skill or topic . Typically offered digitally through bite-sized video lessons or interactive practice exercises, it capitalizes on learners' preference for short-form content and informal learning methods, making knowledge acquisition more accessible and manageable for busy individuals. A defining feature of nano-learning is its brevity, with lessons intentionally kept under two minutes to align with contemporary learning habits, such as engaging with short-form videos on platforms like YouTube Shorts and TikTok . Empirical evidence suggests that the use of short videos is associated with decreased feelings of loneliness and social isolation, thereby reducing depression among older adults . Platforms that allow users to showcase aspects of their own lives also serve as a significant avenue for achieving "happiness in old age" and enhancing social interactions with acquaintances . Therefore, this study aims to provide robust evidence on the effectiveness of nano-learning interventions, particularly in the context of sarcopenia, where addressing physical and psychological well-being has become increasingly critical among this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were 60 years or older,
* had a diagnosis of sarcopenia based on a cut-off score of ≥3 of the Sarcopenia Geriatric Scale (SARCO-GS) (Rosas-Carrasco, 2023),
* able to communicate effectively, and provided informed consent.

Exclusion Criteria:

* Exclusion criteria encompassed severe cognitive impairment, debilitating chronic conditions, or unstable medical status that could hinder participation.
* Cognitive function was assessed using the Montreal Cognitive Assessment (MoCA), with a cutoff score of 25 or below used to exclude participants (Nasreddine, 2005).

Ages: 58 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-07 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
A Composite Physical Function (CPF) Scale | 2 month
  is a validated tool designed to assess functional capacity in older adults across a continuum of daily activities. It consists of 12 items organized hierarchically, beginning with two basic activities of daily living (BADL) related to self-care, eating, and hygiene, followed by eight instrumental activities of daily living (IADL) that assess community functioning such as household chores, shopping, and mobility, and concluded with two advanced activities involving more demanding household tasks and strenuous physical exercise.

SECONDARY OUTCOMES:
Mini Nutritional Assessment-Short Form (MNA-SF) | 2 month
  is a validated screening tool and one of the most widely recognized and well-studied tools for nutritional screening. It is designed to quickly identify older adults who are malnourished or at risk of malnutrition. As a shortened version of the full Mini Nutritional Assessment, it is widely used in clinical, community, and research settings due to its simplicity and time efficiency (Vellas et al., 2006).
Geriatric Depression Scale-Short Form (GDS-SF) | 2 month
  is a 15-item self-report tool designed to evaluate depression and overall well-being in older adults. Respondents indicate how they have felt during the past week by choosing either "Yes" (scored as 1) or "No" (scored as 0). Scores are summed to yield a total ranging from 0 to 15, with 0-4 reflecting no depression, 5-8 indicating mild depression, 9-11 suggesting moderate depression, and 12-15 representing severe depression. In 2013, Elhusseini translated the scale into Arabic, confirming its validity and reliability (r = 0.70). The GDS-SF remains one of the most effective and widely used geriatric-specific screening instruments for detecting depression in older adults (Abd El Fatah et al., 2022; Stone et al., 2019).

CONTACTS AND LOCATIONS:
Overall Officials: rasha eweida, Principal Investigator — Damanhour University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt